CLINICAL TRIAL: NCT00471120
Title: Feasibility Clinical Study: Accuracy of the P2X7 Biomarker in Detection of Endometrial Cancers in Women
Brief Title: Feasibility Study: Accuracy of Biomarker in Detection of Endometrial Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to protocol deficiencies.
Sponsor: Dick Domanik (Industry)
Responsible Party: Sponsor-Investigator, Dick Domanik, Scientist, CytoCore, Inc.
Organization: CytoCore, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13806-CC113
Record Dates: First submitted 2007-05-07; First posted 2007-05-09 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Uterine Cancer; Endometrial Cancer
MeSH Terms: conditions — Uterine Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P2x7 Assay (Experimental): Compare assay results with biopsy
  Interventions: Other: P2x7 assay

INTERVENTIONS:
Other: P2x7 assay — compare P2X7 assay to biopsy

SUMMARY:
This study aims at developing an accurate, simple, and cost-effective method for screening and early detection of uterine cancers

DETAILED DESCRIPTION:
The present study aims at developing an accurate, simple and cost-effective method for screening and early detection of uterine cancers in women using novel inventions and biotechnology methods for collection and assay of uterine cells. Results of P2X7 assays using tissues obtained from women with known uterine cancer and from women with histologically normal endometrium will be compared. These data will also serve as basis for future studies to test the predictive value of the method in population-based studies.

ELIGIBILITY:
Inclusion Criteria:

* women scheduled to undergo hysterectomy
* ages 18 years and older

Exclusion Criteria:

* pregnant women
* students or employees under the direct supervision on the investigators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy potential of the P2X7 (protein and mRNA levels) for the detection of uterine endometrial cancers in women. | Upon review of the assays.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Pinkerton, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (5):
- United States (5):
  - University of Arkansas, Little Rock, Arkansas
  - University Hospital CASE Medical Center, Cleveland, Ohio
  - University of Texas, Dallas, Texas
  - University of Texas, Galveston, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia

REFERENCES:
- [Background] Wang Q, Wang L, Feng YH, Li X, Zeng R, Gorodeski GI. P2X7 receptor-mediated apoptosis of human cervical epithelial cells. Am J Physiol Cell Physiol. 2004 Nov;287(5):C1349-58. doi: 10.1152/ajpcell.00256.2004. Epub 2004 Jul 21. PMID 15269006
- [Background] Wang L, Feng YH, Gorodeski GI. Epidermal growth factor facilitates epinephrine inhibition of P2X7-receptor-mediated pore formation and apoptosis: a novel signaling network. Endocrinology. 2005 Jan;146(1):164-74. doi: 10.1210/en.2004-1026. Epub 2004 Sep 30. PMID 15459114
- [Background] Feng YH, Wang L, Wang Q, Li X, Zeng R, Gorodeski GI. ATP stimulates GRK-3 phosphorylation and beta-arrestin-2-dependent internalization of P2X7 receptor. Am J Physiol Cell Physiol. 2005 Jun;288(6):C1342-56. doi: 10.1152/ajpcell.00315.2004. Epub 2005 Feb 23. PMID 15728711
- [Background] Feng YH, Li X, Wang L, Zhou L, Gorodeski GI. A truncated P2X7 receptor variant (P2X7-j) endogenously expressed in cervical cancer cells antagonizes the full-length P2X7 receptor through hetero-oligomerization. J Biol Chem. 2006 Jun 23;281(25):17228-17237. doi: 10.1074/jbc.M602999200. Epub 2006 Apr 18. PMID 16624800
- [Background] Li X, Zhou L, Feng YH, Abdul-Karim FW, Gorodeski GI. The P2X7 receptor: a novel biomarker of uterine epithelial cancers. Cancer Epidemiol Biomarkers Prev. 2006 Oct;15(10):1906-13. doi: 10.1158/1055-9965.EPI-06-0407. PMID 17035398